CLINICAL TRIAL: NCT01567007
Title: Impact of Different Interventions in Physical Activity Level and Co-morbidities in Women: Randomized, Controlled Study
Brief Title: Change in Physical Activity Levels in Women at Working Place
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: WOMENPED
Record Dates: First submitted 2012-03-13; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Physical Activity; Obesity
Keywords: pedometer; physical activity; workplace
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (No Intervention): session of 15-20 minutes duration. It took place guidelines on physical activity, delivering a manual with general information about physical activity
- Individual counseling (Experimental): Consisting of three sessions within a maximum period of 3 months. We conducted a counseling, aimed at increasing physical activity, aiming to raise steps. Furthermore, we discuss the importance of physical activity, such as overcoming barriers to physical activity and targets agreed between the parties. The pedometer is given along with a diary to record the number of steps and returned in the last session.
  Interventions: Behavioral: individual counseling
- group counseling (Experimental): The counseling was conducted in groups (10-12 individuals) for 6 sessions at weekly intervals, and two sessions with fortnightly. Each session lasts 60 minutes. The advice is aimed at behavioral changes using the following approaches: advantages and disadvantages of behavior change, how to overcome barriers to physical activity, self-monitoring of physical activity by using the pedometer and setting goals (number of steps / day) in the short term and what to do in case of relapse (not accomplish what was represented) besides livings practices.
  Interventions: Behavioral: group counseling
- aerobic training (Experimental): The fitness program is held two times per week with individuals and groups with three sessions lasts for 40 minutes performed on a treadmill
  Interventions: Behavioral: aerobic training

INTERVENTIONS:
Behavioral: individual counseling — Consisting of three sessions within a maximum period of 3 months. We conducted a counseling, aimed at increasing physical activity, aiming to raise at least 2000 steps over the first week of monitoring. Furthermore, we discuss the importance of physical activity, such as overcoming barriers to physical activity and targets agreed between the parties. The pedometer is given along with a diary to record the number of steps and returned in the last session.
  Arms: Individual counseling
Behavioral: group counseling — The counseling was conducted in groups (10-12 individuals) for 6 sessions at weekly intervals, and two sessions with fortnightly. Each session lasts 60 minutes. The advice is aimed at behavioral changes using the following approaches: advantages and disadvantages of behavior change, how to overcome barriers to physical activity, self-monitoring of physical activity by using the pedometer and setting goals (number of steps / day) in the short term and what to do in case of relapse (not accomplish what was represented) besides livings practices. As the GII and the goal is to raise at least 2000 steps daily on average, with the main focus physical activity in leisure time and transport
  Arms: group counseling
Behavioral: aerobic training — The fitness program is held two times per week with individuals and groups with three sessions lasts for 40 minutes performed on a treadmill.
  Arms: aerobic training

SUMMARY:
The purpose of this study is to evaluate the impact of different types of intervention on physical activity level and co-morbidities in women workers aged between 40 and 50 years. Method: A total of 195 sedentary women aged between 40 and 50 years and those who agreed to participate were randomized to one of the following interventions: GI = Control (n = 47), GII = Individual counseling (n = 53), GIII = Counseling group (n = 48); GIV = physical training set (n = 47). Were evaluated: Physical Activity level (steps number evaluated by a pedometer), quality of life (SF-36), body composition (BMI, waist circumference and bioelectrical impedance) and clinical variables (plasma glucose and blood pressure).

DETAILED DESCRIPTION:
Protocols and Randomization of subjects: Subjects were randomized into 4 groups: control group (GI), individual counseling (GII), group counseling (GIII) and aerobic training set (GIV). The protocols of interventions are described in detail below:

GI - Control: Comprising session of 15-20 minutes duration. It took place guidelines on physical activity, delivering a manual with general information about physical activity.

GII - Individual counseling: Consisting of three sessions within a maximum period of 3 months. We conducted a counseling, aimed at increasing physical activity, aiming to raise at least 2000 steps over the first week of monitoring. Furthermore, we discuss the importance of physical activity, such as overcoming barriers to physical activity and targets agreed between the parties. The pedometer is given along with a diary to record the number of steps and returned in the last session.

GIII - Group Counseling: The counseling was conducted in groups (10-12 individuals) for 6 sessions at weekly intervals, and two sessions with fortnightly. Each session lasts 60 minutes. The advice is aimed at behavioral changes using the following approaches: advantages and disadvantages of behavior change, how to overcome barriers to physical activity, self-monitoring of physical activity by using the pedometer and setting goals (number of steps / day) in the short term and what to do in case of relapse (not accomplish what was represented) besides livings practices. As the GII and the goal is to raise steps daily, with the main focus physical activity in leisure time and transport.

GIV - Programmed Aerobic Training: The fitness program is held two times per week with individuals and groups with three sessions lasts for 40 minutes performed on a treadmill.

All interventions lasted between 12 and 15 weeks and were carried out on time or before the commencement of work or during lunch or after work hours.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (no serious chronic disease), sedentary (less than 60 minutes of aerobic physical activity per week scheduled), employees of HC / FMUSP aged between 40 and 50 years.

Exclusion Criteria:

* Perform some type of pharmacotherapy for weight reduction, have a BMI > 45 kg/m2 and have functional limitations that would prohibit the execution of hiking.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Change after 3 and 6 months from Baseline in weekly steps number mean measured by a pedometer | Change after 3 and 6 months of the baseline evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Celso F Carvalho, Phd, Principal Investigator — Universidade de São Paulo, Departamento de Fisioterapia Fonoaudiologia e Terapia Ocupacional
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP - HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ribeiro MA, Martins MA, Carvalho CR. Interventions to increase physical activity in middle-age women at the workplace: a randomized controlled trial. Med Sci Sports Exerc. 2014;46(5):1008-15. doi: 10.1249/MSS.0000000000000190. PMID 24126967